CLINICAL TRIAL: NCT05242848
Title: Integrated Exercise in Opioid Agonist Therapy Clinics: A Randomised Controlled Trial
Brief Title: Integrated Exercise Program in Opioid Agonist Therapy Clinics
Acronym: BAReAktiv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); Helse Vest (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 155386/REK-C
Record Dates: First submitted 2022-02-07; First posted 2022-02-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Substance-Related Disorders
Keywords: Opiate substitution Treatment; Exercise Therapy; Exercise; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention is a supervised group-based exercise intervention for 16 weeks, including two outdoor sessions per week. The workout consists of two parts, endurance and a strength training segment. Every workout follows the same structure and lasts approximately 45 minutes. The exercise starts with roughly 15 minutes of endurance warm-up. After the warm-up follows the interval with eight repetitions of 30 seconds uphill, and the participants can freely choose between walking or running. The desired intensity of the intervals is >13 on Borg-score 20. The session will end with four specific exercises focusing on strength training of large muscle groups, including mm. pectoralis major, rectus abdominis, quadriceps femoris, gluteus maximus and latissimus dorsi. The strength training program follows the same structure as the intervals. Clinical staff, research staff, and people with user experience will supervise the exercise sessions.
Who Masked: Outcomes Assessor
Masking Description: Blinding is regarded as difficult and infeasible. Patients will be informed of the follow-up they will receive, but not on other follow-up alternatives that are used or the exact hypotheses for the study. Outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise intervention (Experimental): The intervention is a supervised group-based exercise intervention for 16 weeks, including two outdoor sessions per week. The workout consists of two parts, endurance and a strength training segment. Every workout follows the same structure and lasts approximately 45 minutes. The exercise starts with roughly 15 minutes of endurance warm-up. After the warm-up follows the interval with eight repetitions of 30 seconds uphill, and the participants can freely choose between walking or running. The desired intensity of the intervals is >13 on Borg-score 20. The session will end with four specific exercises focusing on strength training of large muscle groups, including mm. pectoralis major, rectus abdominis, quadriceps femoris, gluteus maximus and latissimus dorsi. The strength training program follows the same structure as the intervals. Clinical staff, research staff, and people with user experience will supervise the exercise sessions.
  Interventions: Behavioral: Exercise intervention
- Standard (No Intervention): Participants randomised to standard treatment will receive regular OAT clinic follow-up without added supplementation.

INTERVENTIONS:
Behavioral: Exercise intervention — The intervention is a supervised group-based exercise intervention for 16 weeks, including two outdoor sessions per week. The workout consists of two parts, endurance and a strength training segment. Every workout follows the same structure and lasts approximately 45 minutes. The exercise starts with roughly 15 minutes of endurance warm-up. After the warm-up follows the interval with eight repetitions of 30 seconds uphill, and the participants can freely choose between walking or running. The desired intensity of the intervals is >13 on Borg-score 20. The session will end with four specific exercises focusing on strength training of large muscle groups, including mm. pectoralis major, rectus abdominis, quadriceps femoris, gluteus maximus and latissimus dorsi. The strength training program follows the same structure as the intervals. Clinical staff, research staff, and people with user experience will supervise the exercise sessions.
  Arms: Exercise intervention

SUMMARY:
Background: Drug use is associated with unhealthy lifestyle choices, resulting in adverse social and health consequences. Particular people with opioid dependence have high morbidity and reduced quality of life. A reduction in fitness level for people with substance use disorder reduces the general health and quality of life. Physical activity is recommended as an adjunctive treatment for people with substance use disorder. Due to its positive effects on health, quality of life and substance use. There is minimal evidence from well-controlled randomised trials among people receiving opioid agonist therapy. However, studies indicate that exercise could be promising in opioid agonist therapy.

Study design: BAReAktiv is a multicentre randomised controlled trial. The study aims to recruit approximately 225 patients receiving opioid agonist therapy.

Intervention: A 16-week group-based exercise intervention with workouts twice a week. The exercise program will consist of endurance and strength training. The intervention will be integrated into outpatient's clinics in Bergen and Stavanger, Norway.

Study population: The target group will be patients over 18 years of age with severe opioid use disorder receiving OAT in outpatient clinics.

Expected outcome: This study will inform the relative advantages and disadvantages of an integrated exercise program as an adjunctive treatment. Both physical and mental health outcomes are of interest. Further scale-up will be considered if the provided exercise program is safe and effective.

DETAILED DESCRIPTION:
See below each section

ELIGIBILITY:
Inclusion Criteria:

* Receiving OAT from an included outpatient clinic with follow-up weekly
* Low level of physical activity measured using IPAQ (assessed at screening)
* Confirming interest in participating in physical activity intervention and providing informed consent (criteria specified)
* Giving informed consent

Exclusion Criteria:

* Not able to participate in the intervention due to physical disabilities or severe mental disorders
* Being imprisoned or in inpatient treatment settings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Psychological distress | Mid of the intervention period 16 weeks after initiation
  The primary outcome is psychological distress assessed with the Norwegian validated translation ten item version of Hopkins Symptom Checklist (SCL-10) in the mid of the intervention period 16 weeks after initiation (12-20). This will be evaluated with mean SCL-10 item score and compared between intervention and control arm.

SECONDARY OUTCOMES:
Physical functioning | Mid of the intervention period 16 weeks after initiation
  Physical functioning assessed with 4-minutes step-test measuring numbers of steps climbed in period
Physical functioning | Mid of the intervention period 16 weeks after initiation
  Physical functioning assessed using the Norwegian validated translation of the International physical activity questionnaire (IPAQ).
Fatigue Symptom Scale | Mid of the intervention period 16 weeks after initiation
  Changes in fatigue will be assessed with the Fatigue Symptom Scale (FSS-3, 0-18, higher is worse)
Biochemical indicator of inflammation | Mid of the intervention period 16 weeks after initiation
  Biochemical indicators of inflammation measured with C-reactive protein in serum
Health-related quality of life | Mid of the intervention period 16 weeks after initiation
  Changes in quality of life will be assessed with EuroQoL five dimensions (EQ-5D-5L, 0-100, higher is better)

CONTACTS AND LOCATIONS:
Overall Officials: Lars T Fadnes, PHD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - LAR Helse Stavanger HF, Stavanger, Rogaland
  - Department of Addiction Medicine, Haukeland University Hospital, Bergen, Vestland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furulund E, Madebo T, Druckrey-Fiskaaen KT, Vold JH, Nordbotn MH, Dahl E, Dyrstad SM, Lid TG, Fadnes LT; ATLAS4LAR study group. Integrated exercise program in opioid agonist therapy clinics and effect on psychological distress: study protocol for a randomized controlled trial (BAReAktiv). Trials. 2024 Feb 29;25(1):155. doi: 10.1186/s13063-024-07993-2. PMID 38424609
- See also: Related Info — https://helse-bergen.no/avdelinger/rusmedisin/rusmedisin-seksjon-forsking/bar/atlas4lar-kartlegging-og-behandling-av-lungesykdom-i-legemiddelassistert-behandling